CLINICAL TRIAL: NCT00689169
Title: Targeted Intensification by a Preparative Regimen for Patients With High-grade B-Cell Lymphoma Utilizing Standard-dose Yttrium-90 Ibritumomab Tiuxetan (Zevalin) Radioimmunotherapy (RIT) Combined With High-dose BEAM Followed by Autologous Stem Cell Transplantation (ASCT)
Brief Title: Targeted Intensification With ZBEAM and Autologous Stem Cell Transplantation in Patients With High-grade B-Cell Lymphoma
Acronym: ZBEAM2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZBEAM2; 2007-000270-23 (EudraCT Number)
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Lymphoma, Large Cell, Diffuse
Keywords: Lymphoma; Lymphoma Diffuse; B-Cell lymphoma; Aggressive lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Lymphoma, B-Cell | interventions — ibritumomab tiuxetan; Carmustine; Etoposide; Cytarabine; Melphalan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): ZBEAM (Zevalin, BCNU, Etoposide, Aracytine, Melphalan) ASCT Rituximab
  Interventions: Drug: ZBEAM (Zevalin, BCNU, Etoposide, Aracytine, Melphalan); Procedure: ASCT; Drug: Rituximab

INTERVENTIONS:
Drug: ZBEAM (Zevalin, BCNU, Etoposide, Aracytine, Melphalan) — Zevalin 0.4 mCi/kg: D-14 BCNU 300 mg/m² : D-6 Etoposide 100 mg/m²/12h : D-6 D-5 D-4 D-3 Aracytine 200 mg/m²/12h : D-6 D-5 D-4 D-3 Melphalan 140 mg/m²: D-2
Procedure: ASCT — ASCT : D0
Drug: Rituximab — Rituximab 250 mg/m² :D-21 D-14

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of a preparative regimen utilizing standard-dose Yttrium-90 Ibritumomab Tiuxetan (Zevalin) radioimmunotherapy combined with high-dose BEAM followed by ASCT after first line treatment in patients aged from 18 to 65 years with poor prognosis CD 20 Diffuse Large B-Cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 65 years.
* Patient with pathologically proven, high grade B-cell Lymphoma CD 20 positive (WHO classification) :
* Diffuse large B cell lymphoma.
* Adverse prognostic factors IPI>1
* In Complete Remission, or partial response to first line treatment.
* Previously treated with chemotherapy regimen containing rituximab: R CHOP or R ACVBP
* Chemo-sensitive disease
* PET Scan prior transplant
* Eligible for autologous stem cell transplantation
* With a minimum life expectancy of 3 months.
* Negative HIV, HBV and HCV serologies (in the last 4 weeks except after vaccination).
* Having previously signed a written informed consent.

Exclusion Criteria:

* Histological transformation in diffuse large B cell lymphoma, any type of low grade lymphoma
* More than one line of treatment. Prior transplantation. Prior exposure to Zevalin
* Central nervous system or meningeal involvement by lymphoma.
* Contraindication to any drug contained in the chemotherapy regimen.
* Any serious active disease or co-morbid medical condition (according to the investigator's decision and information provided in the IDB).
* Poor renal function (creatinin level up to 2.5 maximum normal level) unless these abnormalities are related to the lymphoma.
* Poor hepatic function (total bilirubin level up to 30 micro mol/l, transaminases up to 2.5 maximum normal level) unless these abnormalities are related to the lymphoma.
* Poor bone marrow reserve as defined by neutrophils less than 1.5 G/l or platelets less than 100 G/l
* Large bone marrow irradiation more than 40percent.
* Bone marrow infiltration
* Lack of sufficient autologous hematopoietic stem cells for transplantation.
* Prior treatment with murine antibodies
* Known hypersensibility to murine antibodies or proteins
* Any history of cancer during the last 5 years, with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.
* Adult patient unable to give informed consent because of intellectual impairment.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-08; Primary Completion 2011-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Event free survival (EFS): events being death from any cause, relapse for complete responders and unconfirmed complete responders, progression during and after treatment and changes of therapy | 2 years

SECONDARY OUTCOMES:
Overall response rate (ORR) (Complete Response CR and Partial Response PR) | 100 days
  100 days after ASCT

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gisselbrecht, MD, Principal Investigator — Lymphoma Study Association; Christophe Fruchart, MD, Principal Investigator — Lymphoma Study Association
Locations (1):
- service d'onco hématologie adultes, hôpital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fruchart C, Tilly H, Morschhauser F, Ghesquieres H, Bouteloup M, Ferme C, Van Den Neste E, Bordessoule D, Bouabdallah R, Delmer A, Casasnovas RO, Ysebaert L, Ciappuccini R, Briere J, Gisselbrecht C. Upfront consolidation combining yttrium-90 ibritumomab tiuxetan and high-dose therapy with stem cell transplantation in poor-risk patients with diffuse large B cell lymphoma. Biol Blood Marrow Transplant. 2014 Dec;20(12):1905-11. doi: 10.1016/j.bbmt.2014.07.024. Epub 2014 Jul 26. PMID 25072780